CLINICAL TRIAL: NCT03502811
Title: A Contemporary, Prospective Study Evaluating Real-world Experience of Performance and Safety for the Next Generation of MitraClip® Devices (EXPAND)
Brief Title: The MitraClip® EXPAND Study of the Next Generation of MitraClip® Devices
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-518
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-12

CONDITIONS: Mitral Valve Regurgitation; Mitral Regurgitation
Keywords: MitraClip; MitraClip NTR; MitraClip XTR; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MitraClip NTR/XTR System: Percutaneous mitral valve repair using the MitraClip NTR and XTR system
  Interventions: Device: MitraClip NTR/XTR System

INTERVENTIONS:
Device: MitraClip NTR/XTR System — Percutaneous mitral valve repair using the MitraClip NTR/XTR system.

SUMMARY:
The MitraClip EXPAND Study (A Contemporary, Prospective Study Evaluating Real-world Experience of Performance and Safety for the Next Generation of MitraClip Devices) is designed to confirm the safety and performance of the MitraClip NTR System and MitraClip XTR System.

DETAILED DESCRIPTION:
The data collected in this study will be used to evaluate device outcomes and characterize trends in patient selection for MitraClip therapy in contemporary real-world use. Moreover, the data will be assessed to identify patient or mitral valve anatomical characteristics that may be most appropriate for these next generation devices.

The MitraClip EXPAND Study will be conducted on commercial MitraClip NTR System and MitraClip XTR System that have received CE Mark and/or FDA approval as required.

Up to 1,000 subjects at a maximum of 60 sites in Europe and the US were initially planned to enroll in the MitraClip EXPAND Study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who give consent for their participation
2. Subjects scheduled to receive the MitraClip per the current approved indications for use
3. Subjects with Symptomatic MR (≥3+)

Exclusion Criteria:

1. Subjects participating in another clinical study that may impact the follow-up or results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients who will undergo commercial procedures with the MitraClip® NTR System and/or MitraClip® XTR System after required approval of the device is obtained.
Sampling Method: Probability Sample
Enrollment: 1041 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Saibal Kar, MD, Principal Investigator — Cedars Sinai, Los Angeles CA; Prof. Francesco Maisano, MD, Principal Investigator — University Hospital, Zürich
Locations (57):
- United States (22):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Scripps Health, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Davis Medical Center, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - JFK Medical Center, West Palm Beach, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Via Christi Regional Medical Center - St. Francis Campus, Kansas City, Kansas
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Atlantic Health System - Morristown Memorial Hospital, Morristown, New Jersey
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - New York University Hospital, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - St. Thomas Hospital, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Germany (18):
  - München Grosshadern, München, Bavaria
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universitat Mainz, Mainz, Rhinela
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Deutsches Herzzentrum Berlin, Berlin
  - Immanuelklinikum Bernau und Herzzentrum Brandenburg, Bernau
  - Medizinische Einrichtungen der Universitat zu Koln, Cologne
  - St.-Johannes-Hospital, Dortmund
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf
  - Klinikum der Justus-Liebig-Universität, Giessen
  - Universitatsmedizin Gottingen Georg-August-Universitat, Göttingen
  - Katholisches Marienkrankenhaus GmbH, Hamburg
  - Klinikum der Ruprecht-Karls-Universität Heidelberg, Heidelberg
  - Klinikum Karlsburg der Klinikgruppe Dr. Guth GmbH & Co. KG., Karlsburg
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Klinikum Rechts Der Isar der Technischen Universitat Munchen, München
  - Niels-Stensen-Kliniken Marienhospital Osnabrück, Osnabrück
  - Universitatsklinikum Ulm, Ulm
- Israel (2):
  - Hadassah - Ein Kerem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
- Italy (5):
  - Ospedale San Raffaele- Cardiac, Milan, Lombard
  - Ospedale San Raffaele, Milan, Lombard
  - Policlinico San Donato, Milan, Lombard
  - Presidio Ospedaliero Ferrarotto Alessi, Catania, Sicily
  - Centro Cardiologico Monzino, Milan
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
  - UMC Utrecht, Utrecht
- Spain (3):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Puerta de Hierro - Hospital Universitario, Madrid
  - HCU Virgen de la Victoria, Málaga
- Switzerland (3):
  - Kantonsspital, Aarau
  - Inselspital - University Hospital of Bern, Bern
  - Universitaets Spital Zuerich, Zurich
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Kar S, von Bardeleben RS, Rottbauer W, Mahoney P, Price MJ, Grasso C, Williams M, Lurz P, Ahmed M, Hausleiter J, Chehab B, Zamorano JL, Asch FM, Maisano F. Contemporary Outcomes Following Transcatheter Edge-to-Edge Repair: 1-Year Results From the EXPAND Study. JACC Cardiovasc Interv. 2023 Mar 13;16(5):589-602. doi: 10.1016/j.jcin.2023.01.010. PMID 36922046
- [Derived] Shuvy M, von Bardeleben RS, Grasso C, Raake P, Lurz P, Zamorano JL, Asch F, Kar S, Maisano F; EXPAND Investigators. Safety and efficacy of MitraClip in acutely ill (NYHA Class IV) patients with mitral regurgitation: Results from the global EXPAND study. ESC Heart Fail. 2023 Apr;10(2):1122-1132. doi: 10.1002/ehf2.14273. Epub 2023 Jan 4. PMID 36599332
- [Derived] Sodhi N, Asch FM, Ruf T, Petrescu A, von Bardeleben RS, Lim DS, Maisano F, Kar S, Price MJ. Clinical Outcomes With Transcatheter Edge-to-Edge Repair in Atrial Functional MR From the EXPAND Study. JACC Cardiovasc Interv. 2022 Sep 12;15(17):1723-1730. doi: 10.1016/j.jcin.2022.07.023. PMID 36075643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1041 subjects attempted MitraClip procedure as of the cut-off date of August 5, 2020.
Pre-assignment Details: A total of 1045 subjects were screened between April 5, 2018 and March 29, 2019, of which 4 subjects did not have any procedure attempted.
Period: Overall Study
Arm/Group | MitraClip NTR/XTR System
Started | 1041
Completed | 722
Not Completed | 319
Not completed — Death | 157
Not completed — Withdrawal by Subject | 105
Not completed — Lost to Follow-up | 26
Not completed — No Visits (Missed) | 31

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who underwent a MitraClip implant.
Arm/Group | MitraClip NTR/XTR System
Number analyzed (Participants) | 1041
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.3 (9.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 571
  Female | 470
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 420
  Germany | 384
  Israel | 19
  United Kingdom | 3
  Spain | 25
  Netherlands | 31
  Switzerland | 39
  Italy | 120
Cardiac Intervention History: Prior Cardiac Surgeries [Count of Participants; unit: Participants] | 294

OUTCOME MEASURES:

1. Primary Outcome: Safety Measure: Number of Participants With Major Adverse Events (MAE)
Description: MAE was defined as a composite of all-cause Death, Myocardial Infarction, Stroke, or non-elective Cardiovascular (CV) surgery for device related complications (CEC adjudicated).
Time Frame: At 30 Days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip NTR/XTR System
Number analyzed (Participants) | 1036
Participants
  All-cause Death (Cardiovascular Death) | 24
  Myocardial Infarction | 0
  Stroke | 8
  Non-elective CV surgeries for device-related complications | 11

2. Primary Outcome: Performance Measure: Number of Participants With Mitral Regurgitation (MR) Reduction to ≤2+
Description: The performance was measured by Mitral Regurgitation (MR) Reduction to ≤2+ at 30-day visits.
Time Frame: At 30 days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip NTR/XTR System
Number analyzed (Participants) | 864
Participants | 845

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MitraClip NTR/XTR System
All-Cause Mortality (participants affected / at risk) | 157/1041
Serious Adverse Events (participants affected / at risk) | 392/1041
Other Adverse Events (participants affected / at risk) | 0/1041
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip NTR/XTR System (N=1041)
ANAEMIAS NONHAEMOLYTIC AND MARROW DEPRESSION (Blood and lymphatic system disorders) | 6 (6)
HAEMOLYSES AND RELATED CONDITIONS (Blood and lymphatic system disorders) | 1 (1)
CARDIAC ARRHYTHMIAS (Cardiac disorders) | 54 (56)
CARDIAC DISORDER SIGNS AND SYMPTOMS (Cardiac disorders) | 1 (1)
CARDIAC VALVE DISORDERS (Cardiac disorders) | 32 (32)
CORONARY ARTERY DISORDERS (Cardiac disorders) | 23 (26)
HEART FAILURES (Cardiac disorders) | 181 (250)
MYOCARDIAL DISORDERS (Cardiac disorders) | 3 (3)
PERICARDIAL DISORDERS (Cardiac disorders) | 4 (4)
CARDIAC AND VASCULAR DISORDERS CONGENITAL (Congenital, familial and genetic disorders) | 3 (3)
GASTROINTESTINAL HAEMORRHAGES NEC (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL SIGNS AND SYMPTOMS (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL STENOSIS AND OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS COMPLICATIONS ASSOCIATED WITH DEVICE (General disorders) | 1 (1)
DEVICE ISSUES (General disorders) | 4 (4)
FATAL OUTCOMES (General disorders) | 32 (32)
GENERAL SYSTEM DISORDERS NEC (General disorders) | 6 (10)
HEPATIC AND HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (1)
INFECTIONS - PATHOGEN UNSPECIFIED (Infections and infestations) | 19 (20)
INJURIES NEC (Injury, poisoning and procedural complications) | 5 (5)
PROCEDURAL RELATED INJURIES AND COMPLICATIONS NEC (Injury, poisoning and procedural complications) | 6 (6)
CARDIAC AND VASCULAR INVESTIGATIONS (Investigations) | 1 (1)
HAEMATOLOGY INVESTIGATIONS (Investigations) | 1 (1)
ELECTROLYTE AND FLUID BALANCE CONDITIONS (Metabolism and nutrition disorders) | 1 (1)
GASTROINTESTINAL NEOPLASMS MALIGNANT AND UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LEUKAEMIAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
LYMPHOMAS NON-HODGKIN'S B-CELL (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MISCELLANEOUS AND SITE UNSPECIFIED NEOPLASMS MALIGNANT AND UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
REPRODUCTIVE NEOPLASMS MALE MALIGNANT AND UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RESPIRATORY AND MEDIASTINAL NEOPLASMS MALIGNANT AND UNSPECIFIED (Metabolism and nutrition disorders) | 2 (2)
CENTRAL NERVOUS SYSTEM VASCULAR DISORDERS (Nervous system disorders) | 23 (25)
ENCEPHALOPATHIES (Nervous system disorders) | 1 (1)
MENTAL IMPAIRMENT DISORDERS (Nervous system disorders) | 1 (1)
NEUROLOGICAL DISORDERS NEC (Nervous system disorders) | 5 (5)
NEPHROPATHIES (Renal and urinary disorders) | 1 (1)
RENAL DISORDERS (Renal and urinary disorders) | 8 (8)
URINARY TRACT SIGNS AND SYMPTOMS (Renal and urinary disorders) | 2 (2)
BRONCHIAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
LOWER RESPIRATORY TRACT DISORDERS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PLEURAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 3 (4)
PULMONARY VASCULAR DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY DISORDERS NEC (Respiratory, thoracic and mediastinal disorders) | 18 (18)
CARDIAC THERAPEUTIC PROCEDURES (Surgical and medical procedures) | 2 (2)
SOFT TISSUE THERAPEUTIC PROCEDURES (Surgical and medical procedures) | 1 (1)
ANEURYSMS AND ARTERY DISSECTIONS (Vascular disorders) | 2 (2)
ARTERIOSCLEROSIS, STENOSIS, VASCULAR INSUFFICIENCY AND NECROSIS (Vascular disorders) | 4 (4)
DECREASED AND NONSPECIFIC BLOOD PRESSURE DISORDERS AND SHOCK (Vascular disorders) | 12 (13)
EMBOLISM AND THROMBOSIS (Vascular disorders) | 2 (2)
VASCULAR DISORDERS NEC (Vascular disorders) | 2 (2)
VASCULAR HAEMORRHAGIC DISORDERS (Vascular disorders) | 37 (38)
VASCULAR HYPERTENSIVE DISORDERS (Vascular disorders) | 2 (2)
VASCULAR INJURIES (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03502811/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT03502811/SAP_001.pdf